CLINICAL TRIAL: NCT01045109
Title: Vitamin D and Prostate Cancer
Brief Title: Vitamin D3 Supplementation in Participants Diagnosed With Early-Stage Prostate Cancer Who Decide to Undergo Active Surveillance Treatment Regimen.
Acronym: D3/PCa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRF #P-06-068; CTO# 101121 (Other: MUSC Hollings Cancer Center); MUSC HR# 17398 (Other: MUSC Institutional Review Board); MUSC CTRC #790 (Other: MUSC Clinical and Translational Research Center)
Record Dates: First submitted 2008-01-02; First posted 2010-01-08 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2010-08

CONDITIONS: Prostate Cancer
Keywords: prostate; cancer; vitamin D3; early stage; active surveillance
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open-label vitamin D3 (Experimental): One arm: open-label receiving vitamin D3 4,000 IU daily
  Interventions: Dietary Supplement: cholecalciferol

INTERVENTIONS:
Dietary Supplement: cholecalciferol — 4,000 I.U. softgel daily orally for 48 weeks
  Other Names: vitamin D3
Dietary Supplement: cholecalciferol — cholecalciferol or vitamin D3 4,000 IU daily for 48 weeks
  Other Names: vitamin D3

SUMMARY:
This clinical trial is aimed at measuring the effect of vitamin D3 supplementation on serum prostate-specific antigen (PSA) levels in patients diagnosed with early stage, low-grade, low-risk prostate cancer (Gleason score less than/equal to 6; PSA less than/equal to 10; clinical stage T1C or T2a), who elect to have their disease monitored through active surveillance for at least one year.

ELIGIBILITY:
Inclusion Criteria:

* lowgrade prostate cancer
* serum PSA less than/equal to 10 ng/ml
* Gleason score less than/equal to 6
* referred from their treating physician with treatment plan of active surveillance for one year
* serum creatinine less than/equal to 2.0 mg/dL
* serum phosphate (measured as phosphorus)greater than 2.3 and less than 4.8 mg/dL
* serum calcium greater than 8.5 and less than 10.5 mg/dL

Exclusion Criteria:

* concurrent malignancy, except non-melanoma skin cancer
* history of sarcoidosis
* history of high dose (greater than 1,000 IU daily) vitamin D3 supplementation
* history of hypercalcemia
* treatment with lithium medication

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Effect of vitamin D3 supplementation on prostate specific antigen levels in patients diagnosed with early stage, low-grade, low-risk prostate cancer. | 48 weeks

SECONDARY OUTCOMES:
Safety of subjects (determined by safety lab values every 8 weeks: serum Creatinine, Ca, Phosphorus, PTH, vit D3; CBC with differential; and urine Ca/Creat ratio) taking vitamin D3 supplementation (4,000 I.U.) daily. | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiano Gattoni-Celli, MD, Principal Investigator — MUSC Department of Radiation Oncology
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Garrett-Mayer E, Wagner CL, Hollis BW, Kindy MS, Gattoni-Celli S. Vitamin D3 supplementation (4000 IU/d for 1 y) eliminates differences in circulating 25-hydroxyvitamin D between African American and white men. Am J Clin Nutr. 2012 Aug;96(2):332-6. doi: 10.3945/ajcn.112.034256. Epub 2012 Jul 3. PMID 22760568
- See also: Research/findings related to vitamin D3 — http://www.vitamindcouncil.org